CLINICAL TRIAL: NCT04014023
Title: A Multi-center, Randomized, Double-Blind, Placebo-controlled, Phase 2, Therapeutic Exploratory Study to Evaluate the Efficacy and Safety of DWP16001 in Patients With Type 2 Diabetes Mellitus
Brief Title: Study to Evaluate the Efficacy and Safety of DWP16001 in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DWP16001201
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Enavogliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DWP16001 Amg (Experimental): DWP16001 Amg, Tablets, Orally, Once daily
  Interventions: Drug: DWP16001; Drug: Placebo
- DWP16001 Bmg (Experimental): DWP16001 Bmg, Tablets, Orally, Once daily
  Interventions: Drug: DWP16001; Drug: Placebo
- DWP16001 Cmg (Experimental): DWP16001 Cmg, Tablets, Orally, Once daily
  Interventions: Drug: DWP16001; Drug: Placebo
- Placebo (Placebo Comparator): Placebo, Tablets, Orally, Once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWP16001 — DWP16001 tablets
  Arms: DWP16001 Amg; DWP16001 Bmg; DWP16001 Cmg
Drug: Placebo — DWP16001 placebo-matching tablets

SUMMARY:
The purpose of this study is to determine the efficacy and safety of DWP16001 compared to placebo in the treatment of type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 80 years
* Patients who was diagnosed with type 2 diabetes mellitus at least 8 weeks before
* Body Mass Index (BMI) between 20 and 45 kg/㎡
* Patients with 7% ≤ HbA1c ≤ 10% at screening
* Subject who has conducted a stable diet and exercise for at least 8 weeks

Exclusion Criteria:

* Type 1 diabetes mellitus or secondary diabetes
* Severe diabetes complications (proliferative diabetic retinopathy, stage 4 or higher nephropathy or severe diabetic neuropathy, diabetic ketoacidosis)
* Clinical significantly renal disorders
* Creatinine clearance < 60ml/min (0.84ml/s/㎡) or Glomerular filtration rate(eGFR) < 60mL/min/1.73
* Severe gastrointestinal disorder
* Uncontrolled hypertension (SBP >180 mmHg or DBP > 110 mmHg)
* History of Acute coronary syndrome, unstable angina, myocardial infarction requiring hospitalization, stroke, transient ischemic attack, severe heart failure (NYHA class III/IV), or heart arrhythmia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | at 12 weeks

SECONDARY OUTCOMES:
Change from baseline in FPG | at week 4, 8, 12
The proportion of patients who achieve HbA1c < 7.0%, HbA1c < 6.5% and HbA1c reduction >0.5% from baseline | at week 4, 8, 12

CONTACTS AND LOCATIONS:
Locations (1):
- Daewoong pharmatceutical, Seoul, South Korea